CLINICAL TRIAL: NCT03993002
Title: Danger Associated Molecular Patterns (DAMP) Mediated Innate Immune Failure and Pneumonia After Trauma - the Harvard-Longwood (HALO) Campus Area Consortium
Brief Title: DAMP-Mediated Innate Immune Failure and Pneumonia After Trauma - the Harvard-Longwood (HALO) Campus Area Consortium
Acronym: HALO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment pause due to COVID-19 exceeded funding period; This is not a suspension of IRB approval.
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Daniel Talmor, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 2016P000144; PR151953 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2018-10-26; First posted 2019-06-20 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Respiratory Failure
Keywords: Mechanical Ventilation; Alevolar stretch; Hyperoxia; Normoxia; Hypercarbia; Normocarbia
MeSH Terms: conditions — Respiratory Insufficiency; Hyperoxia; Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normoxia with Normocarbia (Active Comparator): Mechanical ventilation will be adjusted based on arterial blood gas results. Patient will remain on study settings for 48 hours from achieving target setting. Blood and BAL will be collected at the time of enrollment, at 24 hours, at 48 hours and at 72 hours.
  PaO2 < 100 (FiO2 >= 21%) PaCO2 of 30-40
  Interventions: Other: Normoxia with Normocarbia
- Normoxia with Hypercarbia (Active Comparator): Mechanical ventilation will be adjusted based on arterial blood gas results. Patient will remain on study settings for 48 hours from achieving target setting. Blood and BAL will be collected at the time of enrollment, at 24 hours, at 48 hours and at 72 hours.
  PaO2 < 100 (FiO2 >= 21%) PaCO2 of 50-60
  Interventions: Other: Normoxia with Hypercarbia
- Hyperoxia with Normocarbia (Active Comparator): Mechanical ventilation will be adjusted based on arterial blood gas results. Patient will remain on study settings for 48 hours from achieving target setting. Blood and BAL will be collected at the time of enrollment, at 24 hours, at 48 hours and at 72 hours.
  PaO2 > 250 (FiO2 >= 70%) PaCO2 of 30-40
  Interventions: Other: Hyperoxia with Normocarbia
- Hyperoxia with Hypercarbia (Active Comparator): Mechanical ventilation will be adjusted based on arterial blood gas results. Patient will remain on study settings for 48 hours from achieving target setting. Blood and BAL will be collected at the time of enrollment, at 24 hours, at 48 hours and at 72 hours.
  PaO2 > 250 (FiO2 >= 70%) PaCO2 of 50-60
  Interventions: Other: Hyperoxia with Hypercarbia

INTERVENTIONS:
Other: Normoxia with Normocarbia — PaO2 < 100 (FiO2 >= 21%) PaCO2 of 30-40
  Arms: Normoxia with Normocarbia
Other: Normoxia with Hypercarbia — PaO2 < 100 (FiO2 >= 21%) PaCO2 of 50-60
  Arms: Normoxia with Hypercarbia
Other: Hyperoxia with Normocarbia — PaO2 > 250 (FiO2 >= 70%) PaCO2 of 30-40
  Arms: Hyperoxia with Normocarbia
Other: Hyperoxia with Hypercarbia — PaO2 > 250 (FiO2 >= 70%) PaCO2 of 50-60
  Arms: Hyperoxia with Hypercarbia

SUMMARY:
The mortality burden of trauma in the United States is substantial, and is currently the leading cause of death in warfare and in civilians below age 45. Infection and sepsis are leading causes of morbidity and death in early survivors. Pneumonia (PNA) occurs in 17-36% of ventilated trauma patients; far more than non-trauma patients. The long held dogmatic notion of a mechanical predisposition to development of pneumonia in trauma has lacked robust support. However, there is evidence of the innate immune response to injury plays a major role in increasing susceptibility to infection.

This application is for support of a Focused Program Award addressing the role that "danger signaling" due to "danger associated molecular patterns" (or DAMPs) derived from somatic tissue injuries play in altering innate immune signaling in the lung in ways that predisposes to PNA. This innate immune response plays a pivotal role in the development and progression of lung inflammation. The organization of the Focused Program Award is into six Projects with collaborators from the Departments of Surgery, Medicine and Anesthesiology at Beth Israel Deaconess Medical Center; the Department of Surgery at Brigham and Women's Hospital and the Departments of Biology and Biological Engineering at Massachusetts Institute of Technology.

The human subjects interaction portion of this project is covered in the Human Subjects & Samples Project of the Award, although the information and tissues obtained from this Project will be shared with the other Projects, and the activities planned for those Projects are outlined in this application.

DETAILED DESCRIPTION:
The purpose of the interventional group is to address Aim 3 of this research study. Aim 3 will be accomplished by randomizing eligible patients to normoxic or hyperoxic conditions with normocarbic or hypercarbic blood concentrations through ventilator adjustments per the factorial design. All four groups are considered within the bounds of standard practice for many mechanically ventilated patients. Investigators will exclude patients in whom these settings could be detrimental. The patient will be on the study settings by hour 60 of mechanical ventilation, and these settings will be held for 48 hours from achieving the target partial pressure of oxygen (PaO2) levels. Upon enrollment, an arterial line will be placed if there is not already one in place, and an arterial blood gas (ABG) will be drawn if no ABG has been drawn in the prior 12 hours to enrollment. Over 1-3 hours following ventilator adjustments, several ABGs will be drawn in order to determine the need for additional ventilator adjustments. Foreseeable adjustments include changes to FiO2, respiratory rate, and tidal volume. Once the desired PaO2 level is achieved ("time 0"), investigators will obtain an ABG q12 hours throughout the 48 hour interventional period. After maintaining the ventilator settings for 48 hours, ventilator management will revert to the clinical team. Blood and bronchoalveolar lavage (BAL) will be collected from the patient at time of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Expected to be on Control Mode Ventilation (CMV) for at least 48 hours from the time of screening

Exclusion Criteria:

* Patients presenting with a primary acute neurological disorder
* Patients who are post cardiac arrest
* Known pregnancy
* Concomitant enrollment in HALO as a case (trauma) patient
* Not committed to full ventilator support
* Treating physician refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Inflammatory markers | Change over hours 24, 48 and 72
  ROS production (output is in relative light units per second (RLU/sec)) using luminol-dependent chemiluminescence, measured every 90 sec over the assay time-course of 60 min. Over thirty surface markers on neutrophil subpopulations, including CD10, CD11b, CD15, CD16, CD45, CD66b, CD45, CD274, CD279, and CD88, at various times after trauma will be analyzed using flow cytometry and CyTOF technology. Where indicated, activation of p38/MK2 intracellular signaling pathway will be analyzed by western blotting, and RNA expression profiles of individual cells will be attempted using single-cell RNA sequencing technologies.

SECONDARY OUTCOMES:
Neutrophil activation | Change over hours 24, 48 and 72
  ROS production (output is in relative light units per second (RLU/sec)) using luminol-dependent chemiluminescence, measured every 90 sec over the assay time-course of 60 min. Over thirty surface markers on neutrophil subpopulations, including CD10, CD11b, CD15, CD16, CD45, CD66b, CD45, CD274, CD279, and CD88, at various times after trauma will be analyzed using flow cytometry and CyTOF technology. Where indicated, activation of p38/MK2 intracellular signaling pathway will be analyzed by western blotting, and RNA expression profiles of individual cells will be attempted using single-cell RNA sequencing technologies.
Purine metabolism | Change over hours 24, 48 and 72
  Conversion of adenosine triphosphate (ATP) and adenosine diphosphate (ADP) into adenosine (ADO) in lymphomononuclear cells obtained from the peripheral blood and BAL of trauma patients and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Talmor, MD MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI fully endorses the sharing of final research data to serve important scientific goals, to be done by publication, communications and online data "mixed mode" sets at the respective PI webpage. The PI will aim for the timely release and sharing of final research data from DoDsupported studies that will enable for use by other researchers.
  The rights and privacy of individuals who participate in sponsored research must be protected at all times. Data intended for broader use should be free of identifiers that would permit linkages to individual research participants and variables that could lead to deductive disclosure of the identity of individual subjects. Should any intellectual property arise which requires a patent, the PI will ensure that the technology (materials and data) remains widely available to the research community in accordance with the NIH Principles and Guidelines documented in http://grants.nih.gov/grants/policy/data_sharing/data_sharing_brochure.pdf.
Time Frame: beginning 12 months after and ending 36 months after primary study publication.
Access Criteria: Proposals should be directed to dtalmor@bidmc.harvard.edu. To gain access, data requestors will need to sign a data access agreement and have any necessary ethics board approvals in place.

REFERENCES:
- [Background] Lord JM, Midwinter MJ, Chen YF, Belli A, Brohi K, Kovacs EJ, Koenderman L, Kubes P, Lilford RJ. The systemic immune response to trauma: an overview of pathophysiology and treatment. Lancet. 2014 Oct 18;384(9952):1455-65. doi: 10.1016/S0140-6736(14)60687-5. Epub 2014 Oct 17. PMID 25390327
- [Background] Zhang Q, Raoof M, Chen Y, Sumi Y, Sursal T, Junger W, Brohi K, Itagaki K, Hauser CJ. Circulating mitochondrial DAMPs cause inflammatory responses to injury. Nature. 2010 Mar 4;464(7285):104-7. doi: 10.1038/nature08780. PMID 20203610